CLINICAL TRIAL: NCT02267486
Title: Exploratory Study for the Validity of a Novel Dementia Rating Scale (QUick QUestion Scale) for Alzheimer's Disease Dementia
Brief Title: Exploratory Study for the Validity of QuQu Scale
Acronym: QuQu
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TRIAD1402; UMIN000016394 (Other: UMIN-CTR)
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Alzheimer Dementia
Keywords: Alzheimer Dementia, AD; patients; cognitive
MeSH Terms: conditions — Alzheimer Disease | interventions — Observation

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- Alzheimer Dementia (AD): Patients with dementia caused by Alzheimer's disease
  Interventions: Other: Standard therapy of Alzheimer Dementia (AD)
- Non-dementia: Patients with cognitive concern without dementia
  Interventions: Other: Observation

INTERVENTIONS:
Other: Standard therapy of Alzheimer Dementia (AD)
  Groups: Alzheimer Dementia (AD)
Other: Observation
  Groups: Non-dementia

SUMMARY:
Examine the construct validity, the group discriminant ability, and the inter-rater reliability of a novel dementia rating scale (QuQu scale: QUick QUestion scale) candidate for the evaluation of patients with Alzheimer Dementia (AD)

ELIGIBILITY:
Inclusion Criteria:

1. Alzheimer Dementia (AD) patients and patients with cognitive concern without dementia
2. Written Informed consent by each subject and/or a legal representative, and study informant. If the doctor decides that the patient has no trouble in understanding this study, the written informed consent of a legal representative may be exempted. If not, this study needs a written informed consent by a legal representative and the patient except the case where the consent is hardly obtained due to the progression of the disease.

Exclusion Criteria:

1. patients with other types of dementia (e.g. vascular dementia, Levy body dementia, frontotemporal dementia)
2. patients with other diseases which cause secondary dementia prior to Alzheimer Dementia (AD)
3. patients with other severe neurological disease or psychiatric disorder without Alzheimer Dementia (AD)
4. patients with other medical conditions where the investigators determine that it is inappropriate for the subject of this study (e.g. inappropriate for the evaluation of dementia rating scale)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Alzheimer Dementia (AD), non-dementia
Sampling Method: Non-Probability Sample
Enrollment: 972 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Novel Dementia Rating Scale (QUick QUestion Scale) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Yu Nakamura, Principal Investigator — Kagawa University School of Medicine
Locations (1):
- Kagawa University School of Medicine, Kida-gun, Kagawa-ken, Japan